CLINICAL TRIAL: NCT04167020
Title: Mucle Resilience: Muscular Markers Predictive of Functional Recovery After Femoral Neck Fracture in Orthogeriatrics
Brief Title: Hip Fracture and Muscle Resilience
Acronym: HIPRESM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Université de Technologie de Compiegne (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180486; 2019-A00770-57 (Other: IDRCB)
Record Dates: First submitted 2019-10-25; First posted 2019-11-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Hip Fracture, Post Surgery Recovery, Muscle Resilience
Keywords: Muscle aging; Hip fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: High definition surface electromyography (HD-sEMG) — HD-sEMG data will be collected by Mobita 32® (TMSi) device

SUMMARY:
The aging of the population is a major public health problem, particularly with regard to the quality of life and the maintenance of autonomy.

The fracture of the upper end of the femur (EFSF) is a pathology:

* Frequent, affecting the elderly: in France, 80,000 patients / year, 83% aged ≥ 75 years (DREES, 2011),
* severe, on mortality and autonomy: 40% will not recover their walking capacity earlier than 6 months, 13% of patients > 85 years old walk unaided at 4 months and 11% of patients will be newly admitted to an institution in 6 months after the fracture (UPOG / PSL data).
* and costly: costs related to acute care (excluding prostheses and osteosynthesis equipment), are estimated at € 475 million for health insurance in France.

Currently, despite optimized orthogeriatric management, it is difficult to predict how the individual will respond / recover from acute stress related to the EFSF. Physical resilience is an emerging concept in medicine that defines the dynamic ability of a subject to resist or recover from functional decline as a result of stress or disruption. In this context, developing new approaches to assessing resilience is important, to take into account this resilience specific to each patient in order to develop a personalized functional rehabilitation strategy. The objective of the HIPRESM study is to be able to identify, in elderly patients after an EFSF intervention, the muscular signature associated with good functional recovery (= physical resilience). The goal of the investigators is to develop software that will provide this muscle signature by measuring and analyzing parameters from high-definition surface electromyography (HD-sEMG). This technology is innovative, non-invasive and portable, CE marked but not yet used in clinical routine.

DETAILED DESCRIPTION:
The aging of the population is a major public health problem with its multifactorial impact, quality of life and the maintenance of autonomy.

The upper femoral fracture (UFF) is a common pathology: in France, it concerns nearly 80.000 patients per year, 83% of whom are aged 75 (DREES, 2011).

The UFF is a pathology with serious consequences, on the mortality but also on the functional level, since 40% of the patients will not recover their walking capacity previous to 6 months, only 13% of the patients over 85 years old will walk unaided to 4 months and 11% of patients will be newly admitted to an institution within 6 months of the fracture (UPOG data, 20% for patients with major neurocognitive disorders, 4% for others). In the literature, at least 25% of elderly people will not recover their previous walking ability, especially for transfers, walking and climbing stairs (Alarcon 2011, Arinzon 2010, Visser 2000).

The UFF is an expensive pathology, whose costs related to acute care (excluding prostheses and osteosynthesis equipment), are estimated at € 475 million in health insurance in France.

Currently, despite optimized orthogeriatric management, it is difficult to predict how the individual will respond/recover from acute UFF-related stress. Physical resilience is an emerging concept in medicine, which defines the dynamic ability of a subject to resist or recover from a functional decline due to stress or disruption. In this context, developing new approaches to assess resilience is important, to take into account each patient's specific resilience in order to develop a personalized functional rehabilitation strategy. The objective of the HIPRESM study is to identify, in older patients after a UFF intervention, the muscle signature associated with good functional recovery (= physical resilience). The objective of the investigators is to identify the parameters derived from high definition surface electromyography (HD-sEMG) by developing software that will provide this muscle signature. This technology is innovative, non-invasive and portable, and already CE marked.

Main objective: to identify HD-sEMG parameters, measured during quadriceps extension of the lower limb not affected by surgery, within 7 days post surgery for UFF, associated with functional status without human assistance (SPPB) at day 30.

Main Evaluation Criterion: To investigate the association between the parameters provided by HD-sEMG (32 simultaneous channels; portable device and software, Mobita®) of the rectus femoris and functional status without human assistance measured by the Short Physical Performance Battery (SPPB = walking speed over 4 meters, chair satnds, balance) at 30 days after surgery for FESF.

Secondary objectives: to study the association between parameters from HD-sEMG measured during quadriceps extension of the lower limb not affected by surgery within 7 days post surgery for FESF and :

1. the walking capacity at D30
2. the autonomy at D30
3. the walking speed over 5m at D30
4. the quality of life on D30
5. the evolution of HD-sEMG muscle quality at D30
6. in-hospital mortality and at D30
7. the time required for rehospitalization
8. the average length of stay in Follow-up Care and Rehabilitation and in the orthogeriatric stream

Secondary evaluation criteria:

1. Walking ability without human assistance: autonomous walking, with technical assistance, impossible, at D30
2. Autonomy measured by the ADL scale at D30
3. Walking speed over 5 meters at D30
4. Quality of life assessed by the EQ5D questionnaire at D30
5. HD-sEMG settings at D30
6. Death in hospital and at D30
7. The time required for rehospitalization
8. The average length of stay in rehabilitation and orthogeriatric care

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 70 years old
* Managed by orthogeriatric unit after upper femoral fracture surgery
* Patient informed of the study and who has not objected to his participation.

Exclusion Criteria:

* Patient bedridden before the femoral fracture, with limited autonomy to bed-chair transfers
* Any other associated fracture
* Cutaneous allergy with adhesive plaster
* BMI ≥ 30 kg / m²
* Cognitive disorders preventing the correct execution of the movement

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older patients aged 70 years old and over, hospitalized in orthogeriatics after upper femoral fracture surgery.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
HD-sEMG correlated to SPPB | Day 30
  Identify HD-sEMG parameters and mesured them during quadriceps muscle extension on lower limb not affected by surgery in the 7th days after UFF surgery, associated to functional status without human assistance (SPPB) at Day 30.

SECONDARY OUTCOMES:
Walking ability at Day 30 | Day 30
  3 possible answers: autonom walk=2, with technical assistance=1, impossible=0 a higher score meaning better outcome min value=0, maximum value=2
Patient autonomy at Day 30 | Day 30
  Activities of Daily Living scale (ADL scale) a hiigher score meaning better outcome min value=0, maximum value=6
5 meters Walking speed at Day 30 | Day 30
  Time measurement, in second, to walk 5 meters
Quality of life at Day 30: European Quality of Life-5 Dimensions questionnaire | Day 30
  European Quality of Life-5 Dimensions (EQ5D questionnaire) a lower score meaning better outcome min value=0, maximum value=20
HD-sEMG parameters at Day 30 | Day 30
  High density surface electromyogram signals obtained from rectus femoris muscle:
  * Maximum average amplitude obtained (mV)
  * Average Signal to Noise Ratio (dB)
Intra hospital Mortality | Day 30
  Number of patient death during hospital stay
Rehospitalization delay | Day 30
  days between end of first hospitalization and begining of rehospitalization
Length of stay in rehabilitation care and Orthogeriatric sector | Day 30
  Mean Length of stay

CONTACTS AND LOCATIONS:
Overall Officials: KIYOKA KINUGAWA, MD, PhD, Principal Investigator — APHP
Locations (4):
- France (4):
  - APHP - Charles Foix Hospital, Ivry-sur-Seine
  - APHP - Rotschild, Paris, Île-de-France Region
  - APHP - Saint-Antoine Hospital, Paris, Île-de-France Region
  - APHP - Pitie Salpetriere Hospital - UPOG, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.